CLINICAL TRIAL: NCT04780568
Title: A Phase Ib Study of AZD9291 (Osimertinib) and BC2059 (Tegavivint) as First-Line Therapy in Patients With Metastatic EGFR-Mutant Non-Small Cell Lung Cancer (NSCLC)
Brief Title: Osimertinib and Tegavivint as First-Line Therapy for the Treatment of Metastatic EGFR-Mutant Non-small Cell Lung Cancer
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Responsible Party: Principal Investigator, Regan Memmott, Principal Investigator, Ohio State University Comprehensive Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OSU-20298; NCI-2021-01360 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2021-02-28; First posted 2021-03-03 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Metastatic Lung Non-Small Cell Carcinoma; Stage IV Lung Cancer AJCC v8; Stage IVA Lung Cancer AJCC v8; Stage IVB Lung Cancer AJCC v8
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — osimertinib; Specimen Handling

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (osimertinib, tegavivint) (Experimental): Patients receive osimertinib PO QD on days 1-28 and tegavivint IV on day 1. Treatment repeats every 28 days for 4 cycles in the absence of disease progression or unacceptable toxicity. Patients then receive osimertinib PO QD on days 1-28. Treatment repeats every 28 days for 4 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Osimertinib; Drug: Tegavivint; Procedure: Echocardiography Test; Procedure: Multigated Acquisition Scan; Procedure: Computed Tomography; Procedure: FDG-Positron Emission Tomography; Procedure: Biospecimen Collection

INTERVENTIONS:
Drug: Osimertinib — Given PO
  Other Names: AZD-9291; AZD9291; Mereletinib; Tagrisso
Drug: Tegavivint — Given IV
  Other Names: BC 2059; BC-2059; BC2059; Tegatrabetan
Procedure: Echocardiography Test — Undergo ECHO
  Other Names: EC; Echocardiography; ECHO
Procedure: Multigated Acquisition Scan — Undergo MUGA scan
  Other Names: Blood Pool Scan; Equilibrium Radionuclide Angiography; Gated Blood Pool Imaging; Gated Heart Pool Scan; MUGA; MUGA scan; Multi-Gated Acquisition Scan; Radionuclide Ventriculogram Scan; Radionuclide ventriculography; RNV
Procedure: Computed Tomography — Undergo CT
  Other Names: CAT; CAT scan; Computed Axial Tomography; computerized axial tomography; Computerized Tomography; CT; CT scan; Diagnostic CAT scan
Procedure: FDG-Positron Emission Tomography — Undergo 18F-FDG PET
  Other Names: FDG; FDG-PET; FDG-PET Imaging
Procedure: Biospecimen Collection — Undergo blood and/or tissue sample collection
  Other Names: Biological sample collection; Biospecimen collected; Specimen Collection

SUMMARY:
This phase Ib trial is to find out the best dose, possible benefits and/or side effects of osimertinib and tegavivint as first-line therapy in treating patients with EGFR-mutant non-small cell lung cancer that has spread to other places in the body (metastatic). Osimertinib and tegavivint may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Assess the safety and tolerability of osimertinib (AZD9291) in combination with tegavivint (BC2059) in patients with metastatic EGFR-mutant non-small lung cancer (NSCLC) and determine the recommended phase 2 dose (RP2D).

SECONDARY OBJECTIVES:

I. Determine the objective response rate (ORR) in patients with metastatic EGFR-mutant NSCLC treated with the combination of AZD9291 and BC2059.

II. Determine the progression free survival (PFS) in patients with metastatic EGFR-mutant NSCLC treated with the combination of AZD9291 and BC2059.

III. Determine the duration of response (DOR) in patients with metastatic EGFR-mutant NSCLC treated with the combination of AZD9291 and BC2059.

IV. Determine the overall survival (OS) in patients with metastatic EGFR-mutant NSCLC treated with the combination of AZD9291 and BC2059.

CORRELATIVE/EXPLORATORY OBJECTIVES:

I. Evaluate biomarkers of EGFR, Notch3, and beta-catenin pathway activity in tumor biopsies and blood samples.

II. Assess the pharmacokinetics (PK) of AZD9291 and BC2059 in patients with metastatic EGFR-mutant NSCLC.

III. Assess circulating tumor deoxyribonucleic acid (DNA) (ctDNA) at baseline, following 2 and 4 weeks of treatment to evaluate for clearance, and at time of progression to assess for changes in EGFR mutation status.

IV. Measure response using computed tomography (CT) tumor volumetry and dynamic positron emission tomography (PET)/CT.

V. Identify a gene signature that may be predictive of treatment response or resistance using ribonucleic acid (RNA) sequencing of tumor tissue.

OUTLINE:

Patients receive osimertinib orally (PO) once daily (QD) on days 1-28 of each cycle and tegavivint intravenously (IV) over 4 hours on days 1, 8, 15, and 22 of each cycle. Cycles repeat every 28 days for 4 cycles in the absence of disease progression or unacceptable toxicity. Patients then receive osimertinib PO QD on days 1-28 of each cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients also undergo echocardiography (ECHO) or multigated acquisition (MUGA) scan, CT, fludeoxyglucose F 18 (18F-FDG) positron emission tomography (PET), and blood sample collection throughout the trial. Patients may also undergo tissue sample collection on study.

After completion of study treatment, patients are followed up for 30 or 90 days and then every 12 weeks for 4 years.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 years. Children are excluded from this study because neither dosing nor safety data are currently available for AZD9291 or BC2059 in patients < 18 years of age
* Pathology-confirmed metastatic NSCLC
* A common activating mutation must be present in the EGFR gene, i.e., exon 19 deletion or L858R. The presence of uncommon EGFR mutations, e.g., G719X, S768I, or L861Q are also permitted if they co-occur with a common activating mutation. Mutation status must be determined using a tumor biopsy by local Clinical Laboratory Improvement Act (CLIA)-certified assessment. Mutations identified by blood-based testing can be provided, but must be verified by tumor biopsy
* The presence of a concurrent T790M mutation, while uncommon in patients who are naïve to treatment with EGFR TKIs, is also permitted
* Measurable disease as defined by Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 criteria
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2 (Karnofsky >= 60%)
* The patient must be able to swallow pills
* Life expectancy > 3 months
* Leukocytes >= 3,000/mcL
* Absolute neutrophil count >= 1,500/mcL
* Platelets >= 100,000/mcL
* Hemoglobin >= 90 g/L
* Total bilirubin =< 1.5 x institutional upper limit normal (ULN) and up to 3 mg/dL for patients with Gilbert's
* Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase [SGOT])/alanine aminotransferase ALT (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 x institutional ULN and =< 5 x institutional ULN for patients with liver metastases
* Creatinine within 1.5 x ULN OR glomerular filtration rate (GFR) >= 50 mL/min/1.73 m^2 (measured or calculated by Cockcroft and Gault equation) -confirmation of creatinine clearance is only required for patients with creatinine levels above institutional upper limit of normal
* If evidence of chronic hepatitis B virus (HBV) infection, HBV viral load must be undetectable on suppressive therapy if indicated
* If history of hepatitis C virus (HCV) infection, it must be treated and have an undetectable viral load
* Patients with treated brain metastases are asymptomatic and not requiring ongoing treatment
* Patients with new or progressive brain metastases (active brain metastases) or leptomeningeal disease are eligible if the treating physician determines that immediate central nervous system (CNS)-specific treatment is not required and is unlikely to be required during the first cycle of therapy. Clinical stability on a stable dose of decadron is permitted
* Patients with a prior or concurrent malignancy whose natural history or treatment will not interfere with the safety or efficacy assessment of the investigational drugs are eligible for this trial
* Patients with known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, should have a clinical risk assessment of cardiac function using the New York Heart Association Functional Classification. To be eligible for this trial, patients must be class 2B or better
* Ability to understand and sign a written informed consent document

Exclusion Criteria:

* Prior treatment with an EGFR TKI in any setting
* Patients who have not recovered from adverse events (AEs) due to prior anti-cancer therapy (i.e., have residual toxicities > grade 1), with the exception of alopecia
* Past medical history of interstitial lung disease, drug-induced interstitial lung disease, radiation pneumonitis requiring steroid treatment, or any evidence of clinically active interstitial lung disease
* Patients who are receiving any other investigational agent or immunotherapy within five half-lives of the compound or 3 months, whichever is greater
* Patients with an uncontrolled intercurrent illness
* Patients with psychiatric illness/social situations that would limit compliance with study requirements
* History of allergic reactions attributed to compounds of similar chemical or biologic composition as BC2059 or AZD9291. Patients with hypersensitivity to any of the inactive excipients should also be excluded
* Currently receiving (or unable to stop use prior to receiving the first dose of study treatment) medications or herbal supplements known to be potent inducers of CYP3A4 (wash-out periods vary. All patients must try to avoid concomitant use of any medications, herbal supplements and/or ingestion of foods with known inducer effects on CYP3A4
* Pregnant women are excluded from this study because BC2059 has the potential for teratogenic or abortifacient effects. There is also an unknown but potential risk for AEs in nursing infants secondary to treatment of the mother with AZD9291 or BC2059. Breastfeeding patients will be excluded
* Patients with a significant history of cardiovascular disease (e.g., myocardial infarction [MI], thrombotic or thromboembolic event in the last 6 months)
* Any of the following cardiac criteria:

  * Mean resting corrected QT interval (corrected QT [QTc] using Fredericia's formula [QTcF]) > 470 msec. RR is the time from the interval of 1 QRS complex to the next measured in seconds and is commonly calculated as (60/HR)
  * Any clinically important abnormalities in rhythm, conduction or morphology of resting ECG (e.g., complete left bundle branch block, third degree heart block, second degree heart block)
  * Any factors that increase the risk of QTc prolongation or risk of arrhythmic events such as decompensated heart failure, hypokalemia, congenital long QT syndrome, family history of long QT syndrome or unexplained sudden death under 40 years of age in first degree relatives, or any concomitant medication known to prolong the QT interval
  * Left ventricular ejection fraction (LVEF) < lower limit of normal (LLN) as assessed by either multigated acquisition (MUGA) scan or echocardiogram (ECHO)
* Patients with active malignancies other than NSCLC or patients with prior curatively treated malignancy at high risk of relapse during the study period with the exception of localized squamous or basal cell skin cancers, ductal carcinoma in-situ (DCIS), or indolent cancer currently on observation (i.e. chronic lymphocytic leukemia [CLL] or low-risk prostate cancer)
* Any evidence of severe or uncontrolled systemic disease, including uncontrolled hypertension and active bleeding diatheses, which in the investigator's opinion makes it undesirable for the patient to participate in the trial or which would jeopardize compliance with the protocol, or active infection with human immunodeficiency virus (HIV). Screening for chronic conditions is not required
* Patients who are at risk for impaired absorption of oral medication including, but not limited to, refractory nausea and vomiting, chronic gastrointestinal diseases, inability to swallow the formulated product or previous significant bowel resection that would preclude adequate absorption of AZD9291
* Judgment by the investigator that the patient should not participate in the study if the patient is unlikely to comply with study procedures, restrictions, or requirements
* Involvement in the planning and/or conduct of the study (applies to both investigator staff and/or staff at the study site)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2022-01-18 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2029-07-31 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose | Up to 28 days

SECONDARY OUTCOMES:
Overall response rate (ORR) | Up to 4 years
  Defined as patients with complete or partial response using Response Evaluation Criteria in Solid Tumors (RECIST) version (v)1.1. will be calculated as the proportion of patients who achieve a response to therapy divided by the total number of evaluable patients. An evaluable patient is defined as an eligible patient who has received at least one dose of therapy. All evaluable patients will be included in calculating the ORR for the study along with corresponding 95% binomial confidence intervals (CIs) (assuming that the number of patients who respond is binomially distributed).
Progression free survival | From initiation of therapy to disease progression or death, assessed up to 4 years
  Survival will initially be modeled using Kaplan-Meier methods, resulting in median survival times with 95% CI, assuming sufficient events have occurred.
Duration of response | From objective response to disease progression or death, assessed up to 4 years
Overall survival | From start of treatment until death of any cause, assessed up to 4 years
  Survival will initially be modeled using Kaplan-Meier methods, resulting in median survival times with 95% CI, assuming sufficient events have occurred.

OTHER OUTCOMES:
Tegavivint (BC2059) pharmacokinetics (PK) | On days 1, 2, 5, 8, 15, 16, 19, and 22 of cycle 1 (each cycle is 28 days)
  Assessed by BC2059 drug levels following combination therapy with BC2059 and AZD9291 in patients with metastatic EGFR activating mutation positive non-small cell lung cancer (NSCLC).
Osimertinib (AZD9291) PK | On days 1, 2, 8, 15, 16, and 22 of cycle 1 (each cycle is 28 days)
  Assessed by AZD9291 drug levels following combination therapy with BC2059 and AZD9291 in patients with metastatic EGFR activating mutation positive NSCLC.
Β-catenin pathway activity | Up to 4 years
  Will be evaluated by measuring serum levels of the secreted transcriptional targets, PAI1 and MMP7 pre- and post-treatment. EGFR and Notch3/B-catenin expression, cellular localization, and pathway activity will also be assessed in voluntary serial tumor biopsies using immunohistochemical analysis.
Circulating tumor deoxyribonucleic acid (ctDNA) | Up to 4 years
  Will be assessed pre- and posttreatment to evaluate for clearance, as well as at time of progression to assess for changes in EGFR mutation status.
Fludeoxyglucose F 18 (18F-FDG) positron emission tomography (PET) imaging | Baseline to 4 years
  Assessed by static (standardized uptake value [SUV]max, average SUV, tumor-to-background ratio, metabolic tumor volume, total lesion glycolysis) and dynamic (net influx rate constant and glucose metabolic rate at 30 and 60 minutes) parameters will be assessed in patients with metastatic EGFR activating mutation positive NSCLC. 18F-FDG-PET parameters will also be summarized at baseline and after treatment using mean +/- SEM, range, and median. The changes in the FDG-PET/computed tomography parameter measurements from baseline to after treatment will be compared between responders and non-responders using two sample t-test or Wilcoxon test, whichever is appropriate. Logistics regression model might also be used to identify potential predictive and prognostic biomarkers beyond any genomic alteration with response to study drugs.

CONTACTS AND LOCATIONS:
Overall Officials: Regan M Memmott, M.D., Ph.D, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (1):
- Ohio State University Comprehensive Cancer Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The Jamesline — http://cancer.osu.edu